CLINICAL TRIAL: NCT03190200
Title: MRI Findings of Epiphyseal Growth Plate in Healthy Children
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: ORTHOSURG-2017-25849
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: OCD - Osteochondritis Dissecans
MeSH Terms: conditions — Osteochondritis Dissecans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MRI: Subjects with healthy knees
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — No intervention - observational trial using MRI

SUMMARY:
The purpose of the study is to determine if by using MRI changes can be identified changes early on in the knees of young children that may be at risk for developing osteochondritis dissecans. If MRI can identify changes then better council can be offered about the risks of future activity and treatment options.

DETAILED DESCRIPTION:
Each subject will be asked to undergo an MRI at enrollment, six,12, and 18 months. Subjects will be monitored for evidence of osteochondritis dissecans in order to determine if we can identify it and then create a treatment program to allow these children to avoid developing definitive disease

ELIGIBILITY:
Inclusion Criteria:

6-10-year-old children with a sibling with known OCD and 6-10-year-old children with a known OCD in the contralateral knee

Exclusion Criteria:

Unable to undergo an MRI

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 6-10-year-old children with a sibling with known OCD and 6-10-year-old children with a known OCD in the contralateral knee
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
OCD | 18 months
  The Development of Osteochondritis Dissecans is the outcome of interest

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No